CLINICAL TRIAL: NCT01004016
Title: A Double-blind, Placebo-controlled, Crossover Study, Followed by Open-label Study of KPS-0373 in Patients With SCD
Brief Title: A Study of KPS-0373 in Patients With Spinocerebellar Degeneration (SCD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KPS1202
Record Dates: First submitted 2009-10-27; First posted 2009-10-29 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Spinocerebellar Degeneration
Keywords: Spinocerebellar degeneration; Thyrotropin-Releasing Hormone (TRH); SCD
MeSH Terms: conditions — Spinocerebellar Degenerations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- KPS-0373 (Experimental)
  Interventions: Drug: KPS-0373

INTERVENTIONS:
Drug: KPS-0373
  Arms: KPS-0373
Drug: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of KPS-0373 in patients with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Japanese SCD patients with mild to moderate ataxia

Exclusion Criteria:

* Patients with secondary ataxia
* Patients with clinically significant hepatic, renal, or cardiovascular dysfunction

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)

PRIMARY OUTCOMES:
Scale for Assessment and Rating of Ataxia (SARA) | 4 weeks + 12 weeks
Upper and lower extremity function | 4 weeks + 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiro Omori, Study Director — Clinical Development Department, Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Japan, Japan, Japan